CLINICAL TRIAL: NCT06814626
Title: Role of Nutritional Intervention with Friliver for the Treatment of Sarcopenia in Cirrhotic Patients with Refractory Ascites Candidate to Transjugular Intrahepatic Portosystemic Shunt Placement and Identification of Prognostic Factors Related to Clinical Outcome
Brief Title: Role of Nutritional Intervention for the Treatment of Sarcopenia in Cirrhotic Patients with Refractory Ascites Candidate to Transjugular Intrahepatic Portosystemic Shunt Placement and Identification of Prognostic Factors Related to Clinical Outcome
Acronym: NS-TIPS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRRB/31/20
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Liver Cirrhosis; Refractory Ascites in Patients with Cirrhosis; Sarcopenia in Liver Cirrhosis
Keywords: nutritional treatment; sarcopenia; liver cirrhosis; refractory ascites; transjugular intrahepatic portosystemic shunt placement; TIPS
MeSH Terms: conditions — Liver Cirrhosis; Sarcopenia; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12 weeks post-TIPS nutritional dietary intervention (Experimental)
  Interventions: Dietary Supplement: 12-week nutritional intervention with Friliver dispensing; Other: 12-week nutritional intervention with personalized diet; Other: 12-week nutritional intervention with diet diary to report foods eaten.
- Standard clinical practice: follow-up post-TIPS placement. (No Intervention)

INTERVENTIONS:
Dietary Supplement: 12-week nutritional intervention with Friliver dispensing — After TIPS placement patients of the treatment group receive a 12-week nutritional intervention that includes a personalized diet, Friliver dispensing (Dompé; 2 sachets 3 times a day) and a diet diary to report the quantity and quality of the foods eaten every single day.
  Arms: 12 weeks post-TIPS nutritional dietary intervention
Other: 12-week nutritional intervention with personalized diet — After TIPS placement patients of the treatment group receive a 12-week nutritional intervention that includes a personalized diet, Friliver dispensing (Dompé; 2 sachets 3 times a day) and a diet diary to report the quantity and quality of the foods eaten every single day.
  Arms: 12 weeks post-TIPS nutritional dietary intervention
Other: 12-week nutritional intervention with diet diary to report foods eaten. — After TIPS placement patients of the treatment group receive a 12-week nutritional intervention that includes a personalized diet, Friliver dispensing (Dompé; 2 sachets 3 times a day) and a diet diary to report the quantity and quality of the foods eaten every single day.
  Arms: 12 weeks post-TIPS nutritional dietary intervention

SUMMARY:
The hypothesis is that in patients with cirrhosis and refractory ascites candidate to TIPS, and sarcopenia (identified by a PMA ≤16 cm² at the level of L3), who are at high-risk of 6-month mortality after TIPS placement, a post-TIPS 12 weeks nutritional intervention is associated with improved post-TIPS prognosis.

The primary objective is to evaluate the effect of a post-TIPS 12 weeks nutritional intervention on liver transplant-free six-month survival in sarcopenic candidates to TIPS for refractory ascites in cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* men and women with an age ≥ 18 and ≤ 80 years
* clinical, radiological or histological diagnosis of liver cirrhosis
* diagnosis of RA
* confirmation of sarcopenia defined in CT scan as the sum of the psoas muscle areas measured at the level of the 3rd lumbar vertebra (PMA) ≤16 cm2
* informed consent signed

Exclusion Criteria:

* severe hepatic insufficiency (bilirubin> 5 mg/dl, MELD score> 18, Child-Pugh score> 9)
* Congestive heart failure class ≥2 according to New York Heart Association criteria (NYHA)
* Active coronary heart disease (myocardial infarction within 6 months of the study)
* Severe pulmonary hypertension suspected on echocardiogram (systolic pulmonary arterial pressure [PAPs]> 35 mmHg) and confirmed with right cardiac catheterization (PAPs> 45mmHg)
* Chronic renal failure (creatinine> 3 mg/dl)
* Performance status ≥2 according to the Eastern Cooperative Oncology Group scale (ECOG)
* History of grade III-IV hepatic encephalopathy or West Haven grade I-II hepatic encephalopathy episodes within the last 3 months
* Uncontrolled systemic sepsis
* Presence of Hepatocellular carcinoma
* Complete portal vein thrombosis
* Active bleeding from gastroesophageal varices. Patients with adequately treated gastroesophageal varices can be included in the study (banding ligation, sclerotherapy)
* Diagnosis of extra hepatic neoplasia
* Transplant recipients
* Patients unable or unwilling to comply with the protocol requirements
* Pregnant or lactating women
* Patients unable to autonomously express their consent (incapable patients)
* any other laboratory condition or result that in the opinion of the Principal Investigator, preclude the subject's participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of survival at 6 months after TIPS assessed using Kaplan-Meier curves. The difference between the survival of the two groups (control and treatment) will be calculated using a Log-Rank test. | From enrollment to 6 months after TIPS.

CONTACTS AND LOCATIONS:
Locations (2):
- IRCCS ISMETT - Istituto Mediterraneo per i Trapianti e le Terapie ad Alta Specializzazione, Palermo, Italy
- University Clinic for Visceral Surgery and Medicine, Inselspital, Bern, Switzerland